CLINICAL TRIAL: NCT00377338
Title: Phase II Study of Broncho-Alveoscopy Using Fibered Confocal Fluorescence Microscopy
Brief Title: Safety and Accuracy of Alveoscopy in Interstitial Lung Diseases
Acronym: ALVEOLE
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2005/102/HP; ALVEOLE
Record Dates: First submitted 2006-09-15; First posted 2006-09-18 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Respiratory Tract Diseases
Keywords: Bronchoscopy; Diagnostic imaging; Laser scanning confocal microscopy; Pulmonary Alveoli; Healthy volunteers; Diffuse peripheral lung disease; Focal peripheral lung disease
MeSH Terms: conditions — Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — distal lung biopsy if of tumoral nature (fixed or frozen sample)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Fibered confocal fluorescence microscopy (FCFM), also referred to as Cell-Vizio® (MaunaKea Technologies, France) is a new technique that produces microscopic imaging in a living tissue, through a 1 mm fiberoptic miniprobe that can be introduced into the working channel of the bronchoscope. The system produces real-time imaging of endogenous fluorophores with a 5 µm lateral resolution and a field of view of 600 x 600 µm. FCFM is able to produce dynamic, high-resolution microimaging of the respiratory bronchiolar walls, alveolar ducts and sacs in vivo during endoscopy (a procedure termed as alveoscopy).

The hypothesis of this study is that an alveoscopy makes it possible to analyze the microstructure of the distal airways in vivo and to collect specific morphologic information in patients with interstitial lung diseases.

The goals of this French Phase II trial are:

* to evaluate the tolerance of the alveoscopy
* to describe the normal appearance of the bronchoalveolar system in spontaneous ventilation in normal subjects
* to describe specific alterations of the bronchoalveolar microstructure in focal or diffuse interstitial lung diseases

DETAILED DESCRIPTION:
The study will include 40 healthy smoker or non-smoker volunteers, 20 patients with normal Chest CT scan and normal respiratory function tests, and 90 patients with focal or diffuse peripheral lung diseases.

The Alveoscopy will be performed under local anesthesia, in awake patients during a standard bronchoscopy. The Alveoscopy will be performed on one side of the bronchial tree (left or right lung). Two to ten separate bronchial areas will be explored in each patient, depending on the pathology, focal or diffuse, and the underlying respiratory function.

A continuous monitoring of the Oxygen saturation, blood pressure, EKG will be performed during the procedure. A chest X-ray will be performed after the procedure to eliminate a pneumothorax.

The morphometric parameters of the alveolar microstructure and their variability will be studied according to the age, gender, lung area explored, smoking status in healthy volunteers and "normal CT scan" subjects, as well as in patients with peripheral lung diseases.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers: normal chest X-rays and normal lung function tests
* Patients without parenchymal lung diseases: normal chest computed tomography (CT) scan, normal lung function tests, indication for a bronchoscopy
* Patients with parenchymal lung disease: indication for a bronchoscopy
* Written informed consent for the alveoscopy

Exclusion Criteria:

* Bleeding disorders
* Pulmonary hypertension
* Contraindication for a bronchoscopy
* known hypersensitivity to the fluorescent contrast agent (if required)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy smoker and non-smoker subjects, patients with no peripheral lung disease on CT scan, Patients with focal parenchymal lung diseases, patients with diffuse parenchymal lung diseases
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2006-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
number of lesions localized by confocal endoscopy compared to navigational bronchoscopy | time of the confocal endoscopy compared to navigational bronchoscopy
Positive and negative predictive values of confocal signs before and after IV fluorophore injection for the diagnosis of cancer. | before and after IV fluorophore injection for the diagnosis of cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Luc C Thiberville, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, Haute Normandie, France

REFERENCES:
- [Derived] Salaun M, Guisier F, Dominique S, Genevois A, Jounieaux V, Bergot E, Thill C, Piton N, Thiberville L. In vivo probe-based confocal laser endomicroscopy in chronic interstitial lung diseases: Specific descriptors and correlation with chest CT. Respirology. 2019 Aug;24(8):783-791. doi: 10.1111/resp.13507. Epub 2019 Feb 27. PMID 30811085